CLINICAL TRIAL: NCT03083535
Title: To Evaluate the Efficacy of Aloe Vera Gel in Gingival Massaging and as an Adjunct to Scaling and Root Planing in Patients With Chronic Periodontitis
Brief Title: Efficacy of AloeVera Gel Gum Massaging and Adjunct to Scaling and Root Planing in Chronic Periodontitis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, Neha Mansoriya, Dr., Government College of Dentistry, Indore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCDI
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: CHRONIC PERIODONTITIS
MeSH Terms: conditions — Chronic Periodontitis | interventions — Toothbrushing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tooth Brushing (Active Comparator): Tooth brushing with dentifrice and standardized tooth brush
  Interventions: Procedure: Tooth Brushing
- Aloe vera massaging (Experimental): Tooth brushing with dentifrice and standardized tooth brush followed by massaging with aloe vera gel
  Interventions: Procedure: Tooth Brushing; Procedure: aloe vera Massaging
- SRP with aloe vera massaging (Experimental): Scaling and root planning was done with ultrasonic scalar. It was followed by aloe vera massaging on half arch for 3 minutes daily
  Interventions: Procedure: Tooth Brushing; Procedure: aloe vera Massaging; Procedure: SRP with aloe vera massaging

INTERVENTIONS:
Procedure: Tooth Brushing — Tooth Brushing with Dentifrice Tooth Brushing with Dentifrice (Standard Tooth Brushing technique will be demonstrated by using same type of tooth brush and toothpaste).
Procedure: aloe vera Massaging — Tooth Brushing with Dentifrice (with same type of tooth brush and toothpaste) and massaging with aloe vera gel
  Arms: Aloe vera massaging; SRP with aloe vera massaging
Procedure: SRP with aloe vera massaging — on one side of the arch only Scaling and Root Planing(SRP) to be done, while on the other side, after the Scaling and Root Planing massaging with aloe vera ge; shall be carried out by the patients/subjects
  Arms: SRP with aloe vera massaging

SUMMARY:
Periodontal disease is a multifactorial disease caused by mainly bacterial, genetic, immunologically, and environmental factors. Chronic periodontitis, one of the widely prevalent forms of periodontal disease, is characterized by loss of attachment apparatus of the tooth; it can lead to tooth loss. Many non surgical and surgical approaches have been adapted time and again to prevent, intercept, and to treat the various forms of chronic periodontitis. But, these treatment modalities are not approachable by all individuals, because of the various factors such as: low socioeconomic status, illiteracy, high cost of the treatment, no availability of easy and uncomplicated treatment nearby etc. Considering these factors, we are still in need of preventive, practical, and affordable treatment options specially for the population of underdeveloped and developing countries.

DETAILED DESCRIPTION:
Periodontal disease is universally prevalent. It is a multifactorial disease caused by mainly bacterial, genetic, immunologically, and environmental factors. Chronic periodontitis, one of the widely prevalent forms of periodontal disease, is characterized by loss of attachment apparatus of the tooth; it can lead to tooth loss. Many non surgical and surgical approaches have been adapted time and again to prevent, intercept, and to treat the various forms of chronic periodontitis. But, these treatment modalities are not approachable by all individuals, because of the various factors such as: low socioeconomic status, illiteracy, high cost of the treatment, no availability of easy and uncomplicated treatment nearby etc. Considering these factors, we are still in need of preventive, practical, and affordable treatment options specially for the population of underdeveloped and developing countries.

The use of medicinal plants in the prevention and treatment of the various diseases need not to be over emphasized, as their uses had been advocated in treatises: Sushruta Samhita and Charka Samhita, a long back. Now, it is a demand of time to reread and get the valuable informations for the use of Medical and Dental sciences. These information will be very valuable specially, in context of under developed and developing countries.

One of the herbs -'Aloe Vera' is a very important medicinal plant. The name 'Aloe Vera' is derived from the Arabic Word "Alloeh" meaning "Shining bitter substance," while "Vera" in Latin means "true". Over the years, this plant has been known by a number of names such as 'Wand of heaven', 'Heaven's blessing, and 'the Silent healer'. Plant Aloe Vera is known to us since the ancient time which has stiff grey green lance shaped leave. These leaves hold clear gel in a central mucilaginous pulp. This polysaccharide gel is responsible for beneficial properties of Aloe Vera.1 Aloe Vera gel polysaccharide acemannan has been found to be effective in activating macrophages and resulted in improved wound healing in a rat model. A novel anti-inflammatory compound c -glucosyl chromones has been extracted from the Aloe vera gel. Antibacterial property against gram positive and gram negative bacteria has also been documented.2 Some studies have also shown its antifungal, antiviral, bactericidal, and virucidal activities. A number of investigations have attempted to relate the chemical constituents in the gel to specific biological effects, such as wound healing effect,3 skin hydration effect,4 anti ageing effec,5 anti-inflammatory effect,6 anti bacterial property,2 anti fungal property7, anti viral effect,8 immunomodulating effect,9 anti tumour effect,10 and laxative effect.11 In Dentistry, clinical applications of Aloe Vera have been seen in the treatment of Apthous ulcers, Oral lichen Planus, Alveolar osteitis, and denture adhesive.12 Moreover, several studies have shown the efficacy of Aloe Vera in treating Gingivitis.13 In another study the effect of tooth paste containing high concentration of Aloe Vera, has been observed on the reduction of plaque and gingivitis.14 In underdeveloped and developed countries the application of simple and cost effective approaches are required. Therefore, this study has been planned to evaluate the clinical efficacy of Aloe Vera in moderate to severe form of Generalized Chronic Periodontitis in Indian patients.

Very few studies, which can be counted on fingers, have been conducted worldwide. Hence, this study is being taken to evaluate the Efficacy of Aloe Vera Gel in Gingival Massaging and as an Adjunct to Scaling and Root

ELIGIBILITY:
Inclusion Criteria:

* Cases with moderate to severe form of Generalised Chronic Periodontitis patients of any sex.
* Patients in the age group of 35-65 years, who abide by approved protocol guidelines, and are ready to give written informed consent.

Exclusion Criteria:

* Any known systemic disease which has effects on periodontium such as diabetes etc.
* Patients on anti-inflammatory, antibiotics and perioceutics, since 3 months.
* Patients who have known allergy to material used for the study.
* Pregnant and lactating mothers.
* Patients had undergone any kind of non-surgical and/or surgical periodontal therapy earlier, in past 6 months.
* Tobacco users.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | baseline

SECONDARY OUTCOMES:
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | 1 week
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | 2 week
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | 4 week
Plaque Index (Turesky modification of Quigley Hein Index, 1970) | 6 week
Gingival Index (Loe H and Silness J 1963) | baseline
Gingival Index (Loe H and Silness J 1963) | 1 week
Gingival Index (Loe H and Silness J 1963) | 2 week
Gingival Index (Loe H and Silness J 1963) | 4 week
Gingival Index (Loe H and Silness J 1963) | 6 week
Russell's Periodontal Index (Rusell's A.L, 1956) | baseline
Russell's Periodontal Index (Rusell's A.L, 1956) | 1 week
Russell's Periodontal Index (Rusell's A.L, 1956) | 2 week
Russell's Periodontal Index (Rusell's A.L, 1956) | 4 week
Russell's Periodontal Index (Rusell's A.L, 1956) | 6 week
Periodontal Probing Depth | baseline
Periodontal Probing Depth | 1 week
Periodontal Probing Depth | 2 week
Periodontal Probing Depth | 4 week
Periodontal Probing Depth | 6 week
Clinical Attachment Levels | baseline
Clinical Attachment Levels | 1 week
Clinical Attachment Levels | 2 week
Clinical Attachment Levels | 4 week
Clinical Attachment Levels | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: Dr Subhash Garg, MDS, Study Chair — Govt. College of Dentistry Indore, M.P. India,Indore, M.P, India, 452001

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kumar A, Sunkara MS, Pantareddy I, Sudhakar S. Comparison of Plaque Inhibiting Efficacies of Aloe Vera and Propolis Tooth Gels: A Randomized PCR Study. J Clin Diagn Res. 2015 Sep;9(9):ZC01-3. doi: 10.7860/JCDR/2015/13185.6413. Epub 2015 Sep 1. PMID 26501001
- [Background] Mangaiyarkarasi SP, Manigandan T, Elumalai M, Cholan PK, Kaur RP. Benefits of Aloe vera in dentistry. J Pharm Bioallied Sci. 2015 Apr;7(Suppl 1):S255-9. doi: 10.4103/0975-7406.155943. PMID 26015726